CLINICAL TRIAL: NCT03221595
Title: A Multicenter, Randomized Controlled Trial of Surgical Stabilization of Rib Fractures in Patients With Severe, Non-flail Fracture Patterns
Brief Title: Multicenter RCT of SSRF in Non Flail Patients
Acronym: CWISNONFLAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COMIRB 17-1432
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Rib Fracture Multiple

STUDY DESIGN:
Intervention Model Description: randomized, controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Operative (Experimental): Patients in the operative arm will undergo best medical management, in addition to surgical stabilization of their displaced rib fractures within 72 hours of admission to the hospital.
  Interventions: Device: Operative
- Non-operative (No Intervention): Patients in the non operative arm will undergo best medical management of their displaced rib fractures.

INTERVENTIONS:
Device: Operative — This operation involves reducing and providing rigid fixation of displaced rib fractures with permanent plates or splints
  Other Names: Surgical stabilization of rib fractures, rib plating
  Arms: Operative

SUMMARY:
This study evaluates the efficacy of surgical stabilization of rib fractures, as compared to best medical management, for patients with multiple, displaced rib fractures.

Half of patients will be randomized to surgery (in addition to best medical management), whereas the other half will be randomized to medical therapy only.

The primary outcome will be the subjects overall quality of life measured at two months following injury.

DETAILED DESCRIPTION:
Rib fracture are the most common serious injury following blunt trauma, and occur in approximately 10% of trauma patients [1]. Despite improvements in the care of rib fracture patients, outcomes remain poor and have not changed substantially over the last 15 years [2]. Poor outcomes resulting from serious rib fractures include both acute complications (e.g., pneumonia, prolonged mechanical ventilation, and death) and chronic disability (e.g., pain, dyspnea, and loss of productivity).

Over the last 10 years, surgical stabilization of rib fractures (SSRF) has emerged as a promising technology for the management of patients with severe chest wall injuries [3]. Conceptually, SSRF applies the fundamental orthopedic principles of reduction and fixation to rib fractures, restoring chest wall stability and minimizing pain with respiration, splinting, and secretion accumulation. The advent of muscle-sparring [4] and even minimally-invasive surgical techniques [5], as well as a relatively low complication rate [6], has improved the appeal of this operation.

To date, three randomized clinical trials (RCTs) [7-9] and three meta-analyses of these and other trials [10-12] have limited their scope to patients with flail chest, a specific clinical diagnosis characterized by paradoxical motion of a portion of the chest wall due to fractures of two or more ribs in at least two places. Flail chest represents the most severe form of chest wall injury, with an associated, very high morbidity and mortality. Each of the aforementioned RCTs, as well as multiple prospective, non-randomized investigations [13, 14], have found a benefit to SSRF as compared to best medical management in this patient population. Accordingly, expert consensus statements have recommended this operation in this subset of patients [3, 15].

Based upon the favorable reported efficacy of SSRF in patients with flail chest, many surgeons have broadened indications to patients with severe, non-flail rib fracture patterns, most commonly ≥ 3 severely displaced fractures. Although these injuries differ anatomically from flail chest, many of the same pathophysiologic principles are at work: namely, painful motion at the fracture sites cause respiratory compromise, bony bridging [16], and risk of subsequent non-union, chronic pain, and restrictive lung disease. However, it is not clear if stabilization of these fractures confers the same benefits as in the case of flail chest. This lack of efficacy data has been recognized in recent guidelines, which were unable to recommend SSRF for non-flail fracture patterns pending further data. Furthermore, long term quality of life data for both flail and non-flail fracture patterns managed with SSRF are not available.

The use of SSRF is increasing exponentially. Somewhat alarmingly, nearly one half of the procedures were performed in patients without flail chest [17]. A combination of the favorable results observed for SSRD in flail chest, the increasing prevalence of SSRF for non flail-chest, and the lack of quality evidence to support this operation in this patient population, lead to the design of the current RCT. The objective of this trial is to investigate the efficacy of SSRF, as compared to non-operative management, for hospitalized patients with specific, non-flail, severe rib fractures, and within expert, high volume centers that participate in the Chest Wall Injury Society. The investigators hypothesize that SSRF, as compared to standardized medical management, improves pain control, pulmonary function, risk of complications, and quality of life among patients with severe, non-flail chest fracture patterns.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization with ≥ 3 severely displaced (≥ 50% of rib width) acute rib fractures.
2. Two or more of the following pulmonary physiologic derangements (at the time of consideration for enrollment and after best medical therapy).

   1. Respiratory rate > 20 breaths per minute
   2. Incentive spirometry < 50% predicted (appendix D)
   3. Numeric pain score > 5
   4. Poor cough (as documented by respiratory therapist)
3. Surgery anticipated < 72 hours from injury

Exclusion Criteria:

1. Age < 18 years or ≥ 80 years
2. Flail chest: either radiographic or clinical. Radiographic flail chest is defined on CT chest as ≥ 2 ribs each fractured in ≥ 2 places. Clinical flail is defined as visualization of a segment of chest wall with paradoxical motion on physical exam.
3. Moderate or severe traumatic brain injury (GCS at the time of consideration for enrollment < 12)
4. Intubation
5. Severe pulmonary contusion, defined as Blunt Pulmonary Contusion 18 (BPC18) score > 12 [19].
6. Prior or expected emergency exploratory laparotomy during this admission.
7. Prior or expected emergency thoracotomy during this admission.
8. Prior or expected emergency craniotomy during this admission.
9. Spinal cord injury
10. Pelvic fracture that has required, or is expected to require, operative intervention during this admission.
11. The patient was unable to accomplish activities of daily living independently prior to injury (e.g., dressing, bathing, prepearing meals).
12. Pregnancy.
13. Incarceration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredric M Pieracci, MD MPH, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pieracci FM, Majercik S, Ali-Osman F, Ang D, Doben A, Edwards JG, French B, Gasparri M, Marasco S, Minshall C, Sarani B, Tisol W, VanBoerum DH, White TW. Consensus statement: Surgical stabilization of rib fractures rib fracture colloquium clinical practice guidelines. Injury. 2017 Feb;48(2):307-321. doi: 10.1016/j.injury.2016.11.026. Epub 2016 Nov 27. No abstract available. PMID 27912931

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Operative | Non-Operative
Started | 51 | 59
Completed | 51 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Operative | Non-Operative | Total
Number analyzed (Participants) | 51 | 59 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (15.4) | 53.2 (16.1) | 53.6 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 39 | 43 | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51 | 59 | 110

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Score
Description: Patient self-reported pain score on an 11 point scale scale ranging from 0-10; 0 being "no pain" to 10 "the worst pain imaginable".
Time Frame: Hospital days 1-7, day of discharge (an average of 1 week) and at 2, 4 and 8 weeks following discharge from hospital.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 51 | 59
score on a scale
  Hospital day 1 | 7.5 (2.4) | 7 (2.3)
  Hospital day 2 | 6.3 (2.6) | 6.0 (2.4)
  Hospital day 3 | 5.3 (2.8) | 5.9 (2.1)
  Hospital day 4 | 5.3 (2.8) | 6.1 (2.4)
  Hospital day 5 | 5.0 (2.3) | 5.9 (2)
  Hospital day 6 | 4.7 (2.1) | 5.8 (2.1)
  Hospital day 7 | 4.7 (2.6) | 6.3 (2.3)
  Day of discharge | 4.1 (2.3) | 5.2 (2.4)
  2 week follow-up | 2.9 (2.1) | 4.5 (2.2)
  4 week follow-up | 2.4 (2.4) | 3.3 (2.6)
  8 week follow-up | 1.5 (1.3) | 3.3 (2.7)

2. Secondary Outcome: Length of Stay
Description: Patient length of stay in hospital and/or ICU.
Time Frame: 2 months after injury
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 51 | 59
Days
  Hospital length of stay | 7 [5.5 to 10] | 6 [4 to 11]
  ICU length of stay | 2 [0 to 3] | 2 [0 to 3]

3. Secondary Outcome: Daily Narcotic Use
Description: Total standardized narcotic equivalents per day, which is calculated using an equil-analgesic scale:
  Narcotic Dose Unit Route Hydromorphone 1.5 mg IV Hydromorphone 7.5 mg PO Fentanyl 100 mcg IV Morphine 10 mg IV Morphine 30 mg PO Oxycodone 20 mg PO Hydrocodone 30 mg PO
  *IV, intravenous; mcg, micrograms; mg, milligrams; PO, per oral
Time Frame: Inpatient: occurred daily at 10 AM while the patient was hospitalized. Post-discharge: occurred at outpatient clinic follow-up encounter that occurred at 2, 4, and 8 weeks post discharge.
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 51 | 59
mg morphine equivalents
  Hospital Day 1 | 2.6 [1.3 to 4.5] | 1.6 [0.5 to 2.6]
  Hospital Day 2 | 2.0 [0.8 to 3.3] | 2.0 [1.3 to 2.8]
  Hospital Day 3 | 1.5 [0.8 to 3] | 1.6 [1 to 2.3]
  Hospital Day 4 | 1.5 [0.5 to 3] | 1.5 [0.8 to 2.7]
  Hospital Day 5 | 1.3 [0.6 to 2.3] | 2.3 [1 to 3]
  Hospital Day 6 | 1.3 [0.3 to 2.3] | 2.0 [1 to 3.5]
  Hospital Day 7 | 1.0 [0.5 to 2] | 2.3 [0.8 to 3.8]
  Day of Discharge | 0.5 [0.3 to 1.5] | 0.8 [0.5 to 1.5]
  2 Week Follow-up | 0.5 [0 to 1.3] | 1.2 [0.8 to 3]
  4 Week Follow-up | 0.3 [0 to 0.6] | 1.5 [0 to 2]
  8 Week Follow-up | 0.2 [0 to 0.5] | 0.5 [0.3 to 1.3]

4. Secondary Outcome: Incentive Spirometry
Description: The maximum volume (ml) of inspired air through a handheld device called an incentive spirometer. Best value of 3 attempts is recorded. The value of the inspired volume is normalized for patients age, sex, and height and in measured in the percent predicted for that particular individual.
Time Frame: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: % of predicted ml for age/sex/height
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 51 | 59
% of predicted ml for age/sex/height
  Hosp Day 1 | 39 [21 to 61] | 39.5 [27.5 to 49.5]
  Hosp Day 2 | 40 [23 to 59] | 41.5 [32 to 60]
  Hosp Day 3 | 46 [31 to 65] | 49 [42 to 64]
  Hosp Day 4 | 48.5 [33.5 to 67.5] | 49.5 [42 to 66]
  Hosp Day 5 | 59 [37 to 66] | 51 [42 to 59]
  Hosp Day 6 | 52 [41 to 67] | 49 [41.5 to 60]
  Hosp Day 7 | 55 [45 to 72] | 54 [37 to 70]
  Day of Discharge | 63 [55 to 78] | 61 [49 to 74]
  2 Week Follow-Up | 87 [63 to 100] | 90 [73 to 100]
  4 Week Follow-Up | 100 [68 to 112] | 100 [85 to 113]
  8 Week Follow-Up | 100 [81 to 120.5] | 97.5 [77 to 141]

5. Secondary Outcome: Pulmonary Function Testing
Description: Forced expired volume in 1 second, measured in pulmonary function lab
Time Frame: once, at first follow-up, outpatient, clinic visit, which occurred at 2 weeks post discharge.
Measure: Mean (Standard Deviation); unit: % of predicted ml for age/sex/height
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 51 | 59
% of predicted ml for age/sex/height | 75.5 (17.6) | 75.8 (15.8)

6. Secondary Outcome: Number of Patients With Pneumonia
Description: CDC definition of nosocomial pneumonia
Time Frame: Study participants were followed up to 2 months after index admission date.
Measure: Count of Participants; unit: Participants
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 51 | 59
Participants | 1 | 4

7. Secondary Outcome: Days of Ventilator-dependent Respiratory Failure
Description: Mechanical ventilation for > 24 hours at any time during index hospitalization
Time Frame: Study participants were followed up to 2 months after index admission date.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 51 | 59
Days | 0 [0 to 0] | 0 [0 to 0]

8. Secondary Outcome: Chest Wall Specific Quality of Life Questionnaire
Description: An 8 question, validated quality of life (QoL) questionnaire administered at outpatient, clinic follow-up encounters after discharge from the index admission. Minimum score is 0 and indicates the worst outcome of QoL while maximum score is 55, which indicates the highest outcome of QoL.
Time Frame: 2, 4 and 8 weeks after discharge from the index admission
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 51 | 59
units on a scale
  2 Week Follow-Up | 20.6 (11) | 25.3 (10.1)
  4 Week Follow-Up | 16.9 (10.6) | 22.4 (8.8)
  8 Week Follow-Up | 10.4 (10.9) | 15.7 (8.2)

ADVERSE EVENTS:
Time Frame: 2 months after study participant was discharged from index admission.
Arm/Group | Operative | Non-operative
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/59
Other Adverse Events (participants affected / at risk) | 1/51 | 3/59
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operative (N=51) | Non-operative (N=59)
Local Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Unrelated to study. Non-operative subject developed empyema and subsequently underwent VATS decortication
Systemic Infection (Immune system disorders) | 0 (0) | 1 (1) — Unrelated to study. Subject with developed sepsis, which resolved with IV antibiotics
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) — Unrelated to study. Subject experienced hypovolemia which underperfused the kidneys and cause acute, transient renal injury, which resolved with IV fluid administration
Take back to operating room for bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Unrelated to study. By nature of patients trauma, a small bleeding vessel in the subjects diaphragm was only detected after their rib fixation as it was too small to see at the time of the initial operation. Once detected, bleed was repaired in OR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03221595/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT03221595/ICF_001.pdf